CLINICAL TRIAL: NCT07274774
Title: Systemic Therapy Combined With Stereotactic Body Radiotherapy Versus Systemic Therapy Alone in BCLC Stage C Hepatocellular Carcinoma (SCRATCH): A Prospective, Multicenter, Phase II, Randomized Controlled Trial
Brief Title: SBRT Plus Systemic Therapy vs Systemic Therapy Alone in BCLC C Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinbo Yue, Director of Department Radiation Oncology, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2025-074-02
Record Dates: First submitted 2025-11-22; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma; BCLC Stage C Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; BCLC stage C; metastasis; radiotheraphy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasm Metastasis | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): SBRT + Systemic Therapy
  Interventions: Drug: Systemic therapy; Radiation: Radiotherapy
- Control (Other): Systemic therapy will consist of the continuation of the guideline-recommended systemic treatment received prior to enrollment, in accordance with approved labels and national guidelines.
  Interventions: Drug: Systemic therapy

INTERVENTIONS:
Drug: Systemic therapy — Systemic therapy will consist of the continuation of the guideline-recommended systemic treatment received prior to enrollment, in accordance with approved labels and national guidelines
Radiation: Radiotherapy — portal vein tumor thrombus (PVTT, if present) and/or limited extrahepatic active lesions. For patients presenting with more than 10 lesions at baseline (including extrahepatic metastases with or without portal vein tumor thrombus), a comprehensive FDG-PET/CT reassessment of the whole body is required after 3 months of systemic therapy. Patients who demonstrate ≤10 active lesions at this reassessment may then be considered eligible for SBRT. Dose and fractionation: total dose 25-40 Gy delivered in 5 fractions (5-8 Gy per fraction). Dose selection individualized based on tumor size, location and nearby organ-at-risk constraints; sequential or staged SBRT allowed.
  Arms: Treatment

SUMMARY:
This prospective, multicenter, phase II randomized controlled trial compares the efficacy and safety of SBRT combined with systemic therapy versus systemic therapy alone in BCLC stage C hepatocellular carcinoma (HCC). The primary objective is to compare overall survival (OS) between the two arms. Secondary objectives include progression-free survival (PFS), objective response rate (ORR), quality of life (QoL), and incidence and severity of adverse events (AEs). Eligible patients will be randomized 2:1 to an experimental arm (SBRT + systemic therapy) or control arm (systemic therapy alone). Key inclusion criteria include BCLC C disease, Child-Pugh A-B liver function, ECOG ≤2, measurable disease per RECIST 1.1, and stable intrahepatic disease after initial systemic therapy for ≥3 months when applicable. The trial will also include predefined safety monitoring, QoL assessments (EORTC QLQ-C30 and QLQ-HCC18), and exploratory biomarker analyses.

DETAILED DESCRIPTION:
Background: Hepatocellular carcinoma (HCC) is frequently diagnosed at advanced stages with limited curative options. Systemic therapies (targeted agents and immune checkpoint inhibitors) have improved outcomes in BCLC C patients, but their therapeutic effect is unsatisfactory. SBRT provides precise high-dose local control and may synergize with systemic therapy by enhancing tumor immunogenicity and improving local disease control.

Study design: Prospective, randomized, open-label, multicenter Phase II trial. In the experimental arm, patients will continue the guideline-recommended systemic treatment received prior to enrollment, in accordance with approved labels and national guidelines, combined with SBRT delivered to portal vein tumor thrombus (PVTT, if present) and/or limited extrahepatic metastatic lesions. In the control arm, patients will continue the same guideline-recommended systemic treatment without SBRT.

Endpoints: The primary endpoint is overall survival (OS). Secondary endpoints include progression-free survival (PFS), objective response rate (ORR by RECIST 1.1 and mRECIST), disease control rate (DCR), duration of response (DoR), quality of life (EORTC QLQ-C30 and QLQ-HCC18), and safety (CTCAE v5.0). Exploratory endpoints may include biomarker dynamics (e.g., immune cell infiltration, viral markers) and patterns of progression.

Safety and monitoring: AEs will be collected from consent through 30 days after the last radiotherapy; SAEs will be reported per protocol (including deaths up to 90 days after radiotherapy). Regular imaging and clinical assessments will monitor efficacy and safety. Data management and monitoring will follow GCP.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years.
2. Histologically or clinically diagnosed HCC per national guidelines.
3. BCLC stage C (CNLC IIIA/IIIB), including PVTT and/or extrahepatic metastases amenable to protocol procedures.
4. Child-Pugh class A or B (score ≤7).
5. At least one measurable lesion per RECIST 1.1 (criteria specified).
6. ECOG ≤2.
7. Expected survival ≥6 months.
8. Adequate organ function per protocol thresholds.
9. For experimental arm candidates: active lesion count (when PET-CT used) ≤10.
10. If prior initial systemic therapy given: intrahepatic disease stable ≥3 months.
11. Effective contraception from consent through 1 year after treatment end.
12. Ability to understand and sign consent.

Exclusion Criteria:

1. Second primary malignancy (exceptions apply).
2. Tumor thrombus/metastases judged not amenable to radiotherapy.
3. Prior systemic anticancer therapy for current HCC (prior local therapy permitted per rules).
4. Severe organ dysfunction precluding treatment.
5. Uncontrolled comorbidities (e.g., uncontrolled diabetes, active peptic ulcer, severe cardiopulmonary disease).
6. Active uncontrolled infection or active autoimmune disease requiring systemic therapy.
7. Significant neurologic dysfunction.
8. Pregnant or breastfeeding women; no effective contraception.
9. Known hypersensitivity to planned drugs.
10. Any other condition making participation unsuitable per investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2027-11-10 (Estimated); Study Completion 2028-11-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | subjects will be followed up for a minimum combined accrual + follow-up period of 48 months (24-month enrollment + 24-month follow-up planned)
  Time from date of randomization to date of death from any cause

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 2 years
  Time from randomization to radiographic disease progression per RECIST 1.1/mRECIST or death
Objective Response Rate (ORR) | 2 years
  proportion achieving CR or PR by RECIST 1.1 and mRECIST; assessed at scheduled imaging
Disease Control Rate (DCR) | 2 years
  proportion achieving CR + PR + SD
Duration of Response (DoR) | 2 years
  from first documented CR/PR to progression or death
Quality of Life (QoL) | 3 years
  baseline and every 3 months using EORTC QLQ-C30
Quality of Life (QoL) | 3 years
  baseline and every 3 months using EORTC QLQ-HCC18
Treatment-Related Adverse Events (AEs) | 3 months
  from consent through 30 days after last radiotherapy (Serious Adverse Event reporting up to 90 days post-radiotherapy)

OTHER OUTCOMES:
Patterns of Failure (exploratory) | 2 years
  description of local vs distant progression and subsequent treatments.
Biomarker (exploratory): Hepatitis B Virus DNA Level | 2 years
  Quantitative assessment of HBV DNA in peripheral blood as a marker of viral replication.
Biomarker (exploratory): Alpha-fetoprotein (AFP) Level | 2 years
  Serum AFP concentration measured as a tumor burden indicator.
Biomarker (exploratory): Circulating Tumor DNA (ctDNA) Level | 2 years
  Quantification of tumor-derived DNA fragments in peripheral blood using next-generation sequencing.
Biomarker (exploratory): Peripheral Immune Cell Subsets | 2 years
  Flow cytometry-based analysis of circulating immune cell populations
Biomarker (exploratory): ALBI grade | 2 years
  ALBI grade assessed as indicators of survival

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No